CLINICAL TRIAL: NCT01486693
Title: Clinical Outcomes of Topical Ganciclovir Treatment in Cytomegalovirus Anterior Uveitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201109016RC
Record Dates: First submitted 2011-11-16; First posted 2011-12-06 (Estimated); Last update posted 2011-12-06 (Estimated); Status verified 2011-12

CONDITIONS: Anterior Uveitis
Keywords: cytomegalovirus; uveitis
MeSH Terms: conditions — Uveitis, Anterior; Uveitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study was to evaluate long term efficacy and safety of topical ganciclovir treatment in Cytomegalovirus (CMV) anterior uveitis.

DETAILED DESCRIPTION:
The investigators will enroll 60 patients with positive results of the CMV PCR (polymerase chain reaction) from aqueous humor tapping from January 2006 to June 2011. All the patients (40 men, 20 women) were immunocompetent and diagnosed as symptomatic CMV infection. Their medical records will be reviewed, including demographic data as well as their ophthalmic and medical histories.

The purpose of this study was to evaluate long term efficacy and safety of topical ganciclovir treatment in CMV anterior uveitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with positive results of the CMV PCR (polymerase chain reaction) from aqueous humor tapping. All the patients were immunocompetent and diagnosed as symptomatic CMV infection.

Exclusion Criteria:

* Patients without positive results of the CMV PCR
* Immunocompromised patients with positive results of the CMV PCR

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 40 men, 20 women, aged 40-80 years old
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2011-10; Primary Completion 2011-12 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Anterior chamber inflammation | 4 weeks after starting treatment
  anterior chamber cell grading based on slit lamp microscopy

SECONDARY OUTCOMES:
probability of relapse-free | 2 years after treatment
  Kaplan-Meier curve of relapse-free probability

CONTACTS AND LOCATIONS:
Overall Officials: I-Jong Wang, M.D PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Koizumi N, Suzuki T, Uno T, Chihara H, Shiraishi A, Hara Y, Inatomi T, Sotozono C, Kawasaki S, Yamasaki K, Mochida C, Ohashi Y, Kinoshita S. Cytomegalovirus as an etiologic factor in corneal endotheliitis. Ophthalmology. 2008 Feb;115(2):292-297.e3. doi: 10.1016/j.ophtha.2007.04.053. Epub 2007 Jul 31. PMID 17669498
- [Background] Chee SP, Jap A. Cytomegalovirus anterior uveitis: outcome of treatment. Br J Ophthalmol. 2010 Dec;94(12):1648-52. doi: 10.1136/bjo.2009.167767. Epub 2010 Jun 24. PMID 20576767
- [Background] van Boxtel LA, van der Lelij A, van der Meer J, Los LI. Cytomegalovirus as a cause of anterior uveitis in immunocompetent patients. Ophthalmology. 2007 Jul;114(7):1358-62. doi: 10.1016/j.ophtha.2006.09.035. Epub 2007 Feb 12. PMID 17296229